CLINICAL TRIAL: NCT03328754
Title: Comparative Evaluation of Treatment Effects of PowerScope and Forsus Fixed Functional Appliance in Correction of Class II Malocclusion: A Single Centre Randomised Controlled Trial
Brief Title: Comparative Evaluation of PowerScope and Forsus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rekha ortho
Record Dates: First submitted 2017-10-17; First posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Class II Division 1 Malocclusion
Keywords: Pitchfork; Class II malocclusion; PowerScope
MeSH Terms: conditions — Malocclusion, Angle Class II; Overbite

STUDY DESIGN:
Intervention Model Description: Comparative evaluation of treatment effects of PowerScope and Forsus
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was done with Simple Randomisation method to ensure 1:1 allocation ratio and allocation concealment was achieved with similar looking sealed opaque envelopes. The name of the groups 'Forsus' and 'PowerScope' were written on 13 pieces of paper resulting in total 26 pieces of paper which were folded and shuffled in a box, then taken out and without opening put in 26 opaque envelopes which were then sealed and kept again in the box. The envelopes were shuffled inside the box each time the patient was asked to pick one envelope from the box .The patient was assigned to the group mentioned in the envelope which was opened by the primary investigator who was not involved in data analysis..
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Powerscope (Experimental): Powerscope placed bilaterally for class II correction
  Interventions: Device: Powerscope placed bilaterally for class II correction
- Group 2 Forsus (Experimental): Forsus placed bilaterally for class II correction
  Interventions: Device: Group 2 Forsus

INTERVENTIONS:
Device: Powerscope placed bilaterally for class II correction — Powerscope placed bilaterally for class II correction
  Arms: Group 1 Powerscope
Device: Group 2 Forsus — Forsus placed bilaterally for class II correction
  Arms: Group 2 Forsus

SUMMARY:
The objective of this 2-arm parallel double blinded randomized controlled trial is was to evaluate and compare the treatment effects of PowerScope and Forsus in the treatment of Class II division 1 malocclusion. Patient comfort and operator convenience was also assessed and compared .

DETAILED DESCRIPTION:
INTRODUCTION : Among different dental and skeletal combinations that can create a Class II malocclusion, mandibular retrusion is one of the most common characteristics.In such cases, to stimulate mandibular growth by forward positioning of the mandible, various removable and fixed functional appliances are commonly used to alter the position of mandible during the pubertal growth period.

Stimulation of mandibular growth, distal movement of upper dentition, mesial movement of lower dentition contributes to correction of Class II malocclusion with the use of fixed functional appliances. Of the various fixed functional appliances available to the orthodontist today for the correction of Class II malocclusion are Forsus fatigue resistant device which is the most popular fixed functional appliance6 and the PowerScope which is a recent addition to the armamentarium.

PowerScope is delivered as a one-size-fits-all appliance pre-assembled with attachment nuts for quick and easy chairside application. The appliance is a wire-to-wire installation with attachments placed mesial to the first molar in the maxillary arch and distal to the canine of the mandibular arch. Although there are a few case reports in the literature showing the treatment effects and clinical application of PowerScope, there is not a single study mentioning the effects of PowerScope appliance, which has a different status from other fixed functional appliances due to its special attachment. The purpose of this clinical study was to evaluate the skeletal and dental changes produced by the PowerScope and compare these effects with one of the most commonly used fixed functional appliance the Forsus Fatigue Resistant Device (FRD).

MATERIALS AND METHODS: The present study is a prospective, non-pharmacological, double blind, randomised clinical study conducted in the department of Orthodontics and Dentofacial orthopedics, PGIDS Rohtak.

The study sample consisted of 28 patients, were selected from subjects reporting to the department for fixed orthodontic treatment.

The primary researcher explained the nature of the study to the patients and their parents and their consent was taken. The final sample of 28 patients fulfilling the criteria were randomly divided in two groups: Group 1( PowerScope group) and Group 2 (Forsus group) All subjects in both the treatment groups were treated with MBT 0.022- inch slot preadjusted edgewise appliance (Ortho Organizers, San Marcos, Calif). Both arches were levelled and aligned upto 0.019" ×0.025" stainless steel wires and then the fixed functional appliance as per the group mentioned in the patients envelop was installed.

Lateral cephalometric radiographs were taken before starting fixed functional appliance therepy( T1) immediately (1-3 days) before placement of the fixed functional appliance (T2) and after removal of the fixed functional appliance(T3). All cephalometric radiographs were taken on the same cephalostat.

For evaluation of skeletal and dentoalveolar changes that contributed to the Class II correction, pitchfork analysis was used.

To check patient comfort, all the patients were given a questionnaire. The questionnaire was designed in English and then verbally translated into the patients and parents native language at the installation appointment though all the patients and their parents could read and understand it in English. After the installation all the patients were given the questionnaire and requested to bring it at the next scheduled appointment after filling the required details .

ELIGIBILITY:
Inclusion Criteria:

* Patients in active growth period
* Skeletal Class II malocclusion
* Normal or mildly prognathic maxilla
* Retrognathic mandible.
* Increased overjet, not less than 5 mm.
* Horizontal to average growth pattern
* Positive pretreatment visual treatment objective (VTO).
* Minimum crowding in dental arches.
* Treatment completed without any permanent teeth extracted (excluding third molars).

Exclusion Criteria:

* Subjects with a history of orthodontic treatment
* Anterior open bite
* Severe proclination and crowding of anterior teeth
* Any systemic disease affecting bone and generalgrowth
* Vertical growth pattern
* Patient who fails to follow up or undergo complete treatment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
changes in mandibular length | 12 months
  changes in mandibular length after intervention

SECONDARY OUTCOMES:
Evaluation of Patient comfort | 12 months
  questionnaire for evaluating discomfort during parafunctional activities
Evaluation of Operator Convenience | 12 months
  operator convenience by evaluating time taken for placement of each appliance.

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Sharma, Study Director — PGIDS Rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol